CLINICAL TRIAL: NCT05099120
Title: Establishment of Risk Indicators and Early Warning System for Deterioration of Infected Patients in Real-world Data.
Brief Title: Establishment of Risk Indicators and Early Warning System in Infection Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Jingwen Wang
Record Dates: First submitted 2021-10-11; First posted 2021-10-29 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2021-08

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Serious infections refer to life-threatening infections with a morbidity and mortality rate of up to 50%, and are the main cause of death in critically ill patients, mainly including systemic inflammatory response syndrome, sepsis, infectious shock, or systemic multiple organ dysfunction syndrome. Patients with severe infections have rapid disease development, which can cause disorders of cellular circulation and metabolism and impairment of multi-organ function in the early stage, mostly accompanied by clinical complications, and despite the progress of medical technology and the popularization of antibiotic application, the mortality and disability rate is high, which is a hot spot of clinical research today. Patients with severe infections are exposed to a wide range of medical risk factors, including patient factors (advanced age, frailty, malnutrition, long hospital stay, prolonged bed rest), disease factors (immune deficiency, malignancy, diabetes, renal failure, liver failure), drug factors (long-term use of steroid hormones, chemotherapeutic drugs, NSAIDs, etc.), interventional factors (central venous catheter, recent invasive surgery, hemodialysis, endotracheal intubation or mechanical ventilation, etc.), which bring great challenges to clinical treatment. Therefore, early identification of risk indicators for deterioration of infected patients provides a strategic basis for the medical team to take early warning measures to prevent deterioration and poor prognosis, and to reduce the risk of deterioration of patients, which is also the key to reduce the risk of death of infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with infection

Exclusion Criteria:

* Case information is incomplete
* Do not accept follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We integrated pooled individual patient data of infected patients treated at a single center in China from 1 January 2010 until 31 July 2021.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Among patients with infections admitted to the hospital | 30 days of hospitalization
  primary outcome measure were defined as the death.

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Wang, Study Director — The First Affiliated Hospital of Air Force Medical University